CLINICAL TRIAL: NCT07291206
Title: ARBOspot: Characterization of Arbovirus Specific T Cell Response in Patients by Using Enzyme Linked Immunospot (ELISpot) Assays
Acronym: ARBOspot
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Fausto Baldanti, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: ARBOspot
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-10

CONDITIONS: Arbovirus Infections
Keywords: ELISpot; immune response; serology
MeSH Terms: conditions — Arbovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with suspected or confirmed arbovirus infection
  Interventions: Diagnostic Test: Immunological assays for charactarization of T-cell mediated response; Diagnostic Test: Immunological assays

INTERVENTIONS:
Diagnostic Test: Immunological assays for charactarization of T-cell mediated response — ELISpot assay will be performed for monitoring of T-cell mediated response against arboviruses
Diagnostic Test: Immunological assays — Immunological assays for characterization of T-cell mediated respone against arboviruses will be performed in follow-up

SUMMARY:
Arboviruses (arthropod-borne viruses), are a group of RNA viruses that are transmitted to vertebrate hosts by hematophagous arthropods like mosquitos, ticks, and sandflies [1]. In Italy, arboviruses pose a considerable public health concern because of their potential to infect humans and cause severe emergent or re-emergent diseases. Over the past few decades, arboviruses have already been responsible for epidemic outbreaks in Italy, and travels increase the risk of introducing new species previously confined to tropical and sub-tropical regions [2]. Some arboviral infections, like West Nile Virus (WNV), Toscana Virus (TOSV), Sandfly Fever Sicily Virus (SFSV), Sandfly Fever Naples Virus (SFNV), Usutu Virus (USUV), and tick-borne encephalitis virus (TBEV), are considered endemic in Italy [3]. Others, such as Chikungunya Virus (CHIKV), Dengue Virus (DENV), Zika Virus (ZIKV), Yellow Fever Virus (YFV) and Japanese encephalitis Virus (JEV) are under surveillance since imported infections could lead to local outbreaks and subsequent endemic circulation in Italy. Moreover, the increased global travel and unpredictable climate changes could facilitate the spread of arboviral infections [4]. Adequate diagnostic tests play a crucial role in disease surveillance, identifying potential associations between previous infections and chronic diseases and controlling outbreaks by breaking transmission chains. Furthermore, immunological tests can help predict disease severity in healthy and immunocompromised subjects and identify patients at risk for severe disease during secondary infections.

In parallel with direct molecular diagnosis tests, the development of an immunological test capable of determining specific arbovirus T cell response may be useful for diagnostic as well as for epidemiological and investigative purposes. Furthermore, its development provides a set of initial knowledge on which to base the construction of other immunological tests for future emerging viruses, providing tools to counter new epidemic outbreaks. At the same time, the evaluation of immune response is necessary in order to control and contain the spread of these viruses. In conclusion, the present study aims to investigate immunological responses in patients infected with endemic arboviruses circulating in Italy those that could potentially emerging in the future.

Molecular tests have a reduced detectability window in biological samples, which is why often they are not useful for making a diagnosis. Serological tests can give cross-reactivity phenomena between some arboviruses, making differential diagnosis difficult and often inconclusive. Objective is to assess sensitivity of immunological assays for arboviruses-specific T Cell Response (ARBOspot) in order to use them in combination with conventional diagnostic methods.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years- old and over; all sexes will be eligible for the study;
* Suspected arbovirus infection
* Written informed consent and any required authorization obtained from the participant prior to performing any protocol-related procedures;

Exclusion Criteria:

* Any condition that might compromise safety or interfere with study results.
* All other conditions not present in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with suspected arbovirus infection will be included in the study. All the subjects will be enrolled after signature of informed consent. Follow-up will be performed in case of confirmed arbovirus infection.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Performance of T-cell based assays for arboviruses | from enrolment to up 1 year
  Primary endpoint is to evaluate sensitivity of immunological arboviruses Specific T Cell Response assays (ARBOspot) of patients with confirmed arbovirus infection.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy, Italy